CLINICAL TRIAL: NCT02283814
Title: A Phase-1, Open-label, Drug Interaction Study Between Eslicarbazepine Acetate 1200 mg and Topiramate 200 mg Following Multiple Dose Administrations in Healthy Male
Brief Title: A Open-label, Drug Interaction Study Between Eslicarbazepine Acetate and Topiramate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-120
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate; Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A BIA 2-093 + Topamax (Experimental): Group A
  * Pre-treatment: 600 mg once daily dose of eslicarbazepine acetate (ESL) administered for two consecutive days;
  * Treatment 1: 1200 mg once daily dose of eslicarbazepine acetate (ESL) administered for six consecutive days
  * Treatment 2: Concomitant doses of eslicarbazepine acetate (ESL) 1200 mg and TPM 100 mg for two consecutive days
  * Treatment 3: Concomitant doses of eslicarbazepine acetate (ESL) 1200 mg and TPM 100 mg (morning) + 100mg (evening) for two consecutive days
  * Treatment 4: Concomitant doses of eslicarbazepine acetate (ESL) 1200 mg and TPM 200 mg for fifteen consecutive days
  Interventions: Drug: BIA 2-093; Drug: Topamax
- Group B BIA 2-093 + Topamax (Experimental): * Pre-treatment: 100 mg once daily dose of TPM administered for two consecutive days;
  * Pre-treatment 2: 100 mg twice daily dose of TPM administered for two consecutive days;
  * Treatment: 200 mg once daily dose of TPM administered for four consecutive days;
  * Treatment 2: Concomitant doses of eslicarbazepine acetate (ESL) 600 mg and TPM 200 mg for two consecutive days
  * Treatment 3: Concomitant doses of eslicarbazepine acetate (ESL) 1200 mg and TPM 200mg for seventeen consecutive days
  Interventions: Drug: BIA 2-093; Drug: Topamax

INTERVENTIONS:
Drug: BIA 2-093
  Other Names: ESL, Eslicarbazepine acetate
Drug: Topamax
  Other Names: TPM

SUMMARY:
Single centre, open-label, multiple doses, one-sequence design study in two parallel groups of healthy volunteers

DETAILED DESCRIPTION:
Single centre, open-label, multiple doses, one-sequence design study in two parallel groups of healthy volunteers: Group A: Pre-treatment with ESL, treatment with ESL and ascending doses of Topamax (TPM) in last phases; Group B: Pre-treatment with TPM, treatment with TPM and ascending doses of ESL in last phases

ELIGIBILITY:
Inclusion Criteria:

* Availability of volunteer for the entire study period and willingness to adhere to protocol requirements as evidenced by the informed consent form (ICF) duly read, signed and dated by the volunteer
* Male aged of at least 18 years but not older than 45 years with a body mass índex (BMI) greater than or equal to 19 and below 30 kg/m
* Clinical laboratory values within the laboratory's stated normal range; i f not within this range, they must be without any clinical significance (laboratory tests are presented in section 6.1.1.3)
* Healthy according to the medical history, laboratory results and physical
* Light-, non- or ex-smokers. A light smoker is defined as someone smoking 1 0 cigarettes or less per day, and an ex-smoker i s defined as someone who completely stopped smoking for at least 1 2 months before day 1 of this study

Exclusion Criteria:

* Significant history of hypersensitivity to topiramate, eslicarbazepine, oxcarbazepine, carbamazepine or any related products (including excipients of the formulations) as wel l as severe hypersensitivity reactions (like angioedema) to any drugs
* Presence of significant gastrointestinal, l iver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects
* History of significant gastrointestinal, liver o r kidney disease, o r surgery that may affect drug bioavailability, including but not limited to cholecystectomy
* Presence of significant cardiovascular, pulmonary, hematologic, neurologic, psychiatric, endocrine, immunologic or dermatologic d isease
* Presence o f significant heart disease o r disorder according to ECG
* Presence or history of significant central nervous system disorder l ike convulsion or depression
* Presence o r history o f significant ocular disease
* Presence or history of severe hepatic impairment
* Presence or history of renal insufficiency (serum creatinine level greater than 135 μmol/L)
* History or presence of acidosis
* Use of valproic acid in the previous 7 days prior to Day 1 of the study.
* Maintenance therapy with any drug, or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
* Any clinically significant illness in the previous 28 days before day 1 of this study
* Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin and rifampin), in the previous 28 days before Day 1 of this study
* Participation in another clinical trial or donation of 50 mL or more of blood in the previous 28 days before day 1 of this study
* Donation of 500 mL or more of blood (Canadian B lood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before day 1 of this study
* Positive urine screening of drugs of abuse (drugs listing is presented in section 6.1.1.4).
* Positive results to HIV, HBsAg or anti-HCV tests

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-01; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A BIA 2-093 + Topamax: Group A
  * Pre-treatment: 600 mg once daily dose of eslicarbazepine acetate (ESL) administered for two consecutive days;
  * Treatment 1: 1200 mg once daily dose of eslicarbazepine acetate (ESL) administered for six consecutive days
  * Treatment 2: Concomitant doses of eslicarbazepine acetate (ESL) 1200 mg and TPM 100 mg for two consecutive days
  * Treatment 3: Concomitant doses of eslicarbazepine acetate (ESL) 1200 mg and TPM 100 mg (morning) + 100mg (evening) for two consecutive days
  * Treatment 4: Concomitant doses of eslicarbazepine acetate (ESL) 1200 mg and TPM 200 mg for fifteen consecutive days
  BIA 2-093
  Topamax
- Group B BIA 2-093 + Topamax: * Pre-treatment: 100 mg once daily dose of TPM administered for two consecutive days;
  * Pre-treatment 2: 100 mg twice daily dose of TPM administered for two consecutive days;
  * Treatment: 200 mg once daily dose of TPM administered for four consecutive days;
  * Treatment 2: Concomitant doses of eslicarbazepine acetate (ESL) 600 mg and TPM 200 mg for two consecutive days
  * Treatment 3: Concomitant doses of eslicarbazepine acetate (ESL) 1200 mg and TPM 200mg for seventeen consecutive days
  BIA 2-093
  Topamax
Period: Overall Study
Arm/Group | Group A BIA 2-093 + Topamax | Group B BIA 2-093 + Topamax
Started | 16 | 16
Completed | 13 | 14
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A BIA 2-093 + Topamax | Group B BIA 2-093 + Topamax | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Cmax - the Maximum Plasma Concentration
Description: BIA 2-194 and BIA 2-195 are metabolites of eslicarbazepine acetate
Time Frame: Time Frame: Group A:Day 8 and 27: within 5 minutes prior to dosing and 0.5,1,1.5,2,2.5,3,3.5,4,6,9,12,16 and 24 hours after drug administration; Group B: Day 8 and 27 within 5 minutes prior dosing and 0.25,0.5,0.75,1,1.33,1.67,2,2.5,3,4,6,9,12,16 and 24h
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- BIA 2-093 + TPM: BIA 2-093 - ESL; Eslicarbazepine acetate TPM - Topamax
- BIA 2-093: BIA 2-093 - ESL; Eslicarbazepine acetate
Arm/Group | BIA 2-093 + TPM | BIA 2-093
Number analyzed (Participants) | 27 | 16
ng/mL
  Cmax (BIA 2-194) | 21960.6 (2482) | 25414.8 (3736)
  Cmax (BIA 2-195) | 931.8 (216) | 1062.6 (235)

2. Primary Outcome: Tmax - the Time of Occurrence of Cmax
Description: BIA 2-194 and BIA 2-195 are metabolites of eslicarbazepine acetate Both Groups A and B described in participant flow recieved BIA 2-093 and Topiramate. The results presented here are related with the different interventions in both groups
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BIA 2-093 + TPM | BIA 2-093
Number analyzed (Participants) | 27 | 16
hours
  Tmax (BIA 2-194) | 2.00 (0.96) | 2.00 (0.97)
  Tmax (BIA 2-195) | 9.00 (4.20) | 6.00 (3.91)

3. Secondary Outcome: AUCτ - Cumulative Area Under the Plasma Concentration Time Curve Over the Dosing Interval at Steady State.
Description: BIA 2-194 and BIA 2-195 are metabolites of eslicarbazepine acetate
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | BIA 2-093 + TPM | BIA 2-093
Number analyzed (Participants) | 27 | 16
ng*h/mL
  AUCτ (BIA 2-194) | 361733.9 (38706) | 389794.3 (35861)
  AUCτ (BIA 2-195) | 19611.8 (4707) | 22886.8 (5195)

ADVERSE EVENTS:
Arm/Group | Group A BIA 2-093 + Topamax | Group B BIA 2-093 + Topamax
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 15/16 | 13/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A BIA 2-093 + Topamax (N=16) | Group B BIA 2-093 + Topamax (N=16)
Palpitations (Cardiac disorders) | 1 | 0
dry eye (Eye disorders) | 1 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 7
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 4 | 2
Diarrheoa (Gastrointestinal disorders) | 1 | 2
Flatulence (Gastrointestinal disorders) | 2 | 3
hypoaesthesia teeth (Gastrointestinal disorders) | 1 | 0
Lip dry (Gastrointestinal disorders) | 5 | 6
Reflux gastritis (Gastrointestinal disorders) | 1 | 0
Tongue coated (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 5 | 6
Feeling drunk (General disorders) | 2 | 0
Feeling hot (General disorders) | 2 | 0
hot flush (General disorders) | 3 | 1
Pyrexia (General disorders) | 1 | 0
Venipuncture site redness (General disorders) | 1 | 0
Vessel puncture site bruise (General disorders) | 2 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 3
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Red blood cells urine positive (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Arthalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 0
Coordination abnormal (Nervous system disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 4 | 1
Dizziness (Nervous system disorders) | 5 | 1
Headache (Nervous system disorders) | 7 | 4
Somnolence (Nervous system disorders) | 14 | 13
Dysarthria (Nervous system disorders) | 1 | 0
Head discomfort (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 4
Paraesthesia oral (Nervous system disorders) | 8 | 3
Speech disorder (Nervous system disorders) | 1 | 0
Vision blurred (Nervous system disorders) | 1 | 4
Erection increased (Psychiatric disorders) | 1 | 1
Euphoric mood (Psychiatric disorders) | 4 | 3
Irritability (Psychiatric disorders) | 1 | 0
Libido increased (Psychiatric disorders) | 1 | 0
Mood altered (Psychiatric disorders) | 2 | 1
Psychomotor retardation (Psychiatric disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Upper repiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Viral upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 0 | 2
Visual disturbance (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 3
Oral pain (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Blood pressure systolic increased (Investigations) | 0 | 2
Muscular discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1
Coordination decreased (Nervous system disorders) | 0 | 1
Insomnia (Nervous system disorders) | 0 | 1
Sensing disturbance (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Urine abnormality (Renal and urinary disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other